CLINICAL TRIAL: NCT03405415
Title: Assessment of Glucose Concentrations in People Without Diabetes Mellitus After Standardized Meals and in Daily Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IDT-1623-IU
Record Dates: First submitted 2018-01-12; First posted 2018-01-23 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Subjects Without Diabetes Mellitus; Assessment of Glucose Concentrations

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Blood glucose monitoring system and continuous interstitial glucose monitoring system — At enrolment, participants are provided with BGM (Blood Glucose Monitoring) and CGM (Continuous Glucose Monitoring) systems. They will use the systems throughout the study. Participants will visit the study site three times. During the first visit, a standardized oral glucose tolerance test will be performed to ensure that participants do not have diabetes mellitus and to obtain glucose concentration data from people without diabetes mellitus during a glucose challenge. On another two days, participants will visit the study site for standardized breakfast and lunch meals to provide glucose concentration data under standardized conditions.
  Outside of the study site visits, participants are asked to eat similar meals on two days to obtain glucose concentration data under repeated conditions that represent daily life.
  During the study, participants are asked to document meals, physical activity and addition comments to provide context to the recorded glucose concentration data.

SUMMARY:
Participants will perform blood glucose monitoring (BGM) over the course of 14 days and, in parallel, wear continuous glucose monitoring (CGM) systems. Because current CGM systems typically achieve a lower level of analytical accuracy than BGM systems, participants will perform at least 5 blood glucose (BG) measurements per day. In addition, CGM systems are used to obtain minimally-invasive high-frequency glucose measurements to fill the gaps between BG measurements.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Written informed consent
* Subject is legally competent and has the capacity to understand character, meaning and consequences of the study
* Subject is willing to refrain from intake of salicylic acid and ascorbic acid and medication and/or compounds containing these substances

Exclusion Criteria:

* Anamnestically known diabetes mellitus
* Severe acute or chronic disease with potential risk of being adversely affected by the study procedures (at the study physician's discretion)
* Current constitution that compromises the subject's capability to participate in the study (at the study physician's discretion)
* Pregnancy or lactation period
* Known severe skin reactions to adhesives
* Blood donation within the previous two months (according to the subject's statement)
* Language or other barriers potentially compromising an adequate compliance with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-01-27 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
Assessment of glucose concentrations | 14 days per subject

CONTACTS AND LOCATIONS:
Overall Officials: Guido Freckmann, MD, Principal Investigator — Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm
Locations (1):
- Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm, Ulm, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Freckmann G, Schauer S, Beltzer A, Waldenmaier D, Buck S, Baumstark A, Jendrike N, Link M, Zschornack E, Haug C, Pleus S. Continuous Glucose Profiles in Healthy People With Fixed Meal Times and Under Everyday Life Conditions. J Diabetes Sci Technol. 2024 Mar;18(2):407-413. doi: 10.1177/19322968221113341. Epub 2022 Jul 25. PMID 35876145